CLINICAL TRIAL: NCT00309374
Title: Anti-Inflammatory Effect of Statins in the Human Endotoxin Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EK291/2005Version2.0
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Endotoxemia
Keywords: LPS; Statins; leukocyte mRNA expression profiles
MeSH Terms: conditions — Endotoxemia | interventions — Lipopolysaccharides

INTERVENTIONS:
Drug: LPS 2ng/kg intravenous bolus
Drug: Simvastatin 80mg; administered daily p.o. over 5 days
Drug: Rosuvastatin 40mg; administered daily p.o. over 5 days

SUMMARY:
The purpose of this study is to determine the effects of HMG-CoA reductase inhibitor pretreatment on inflammation and coagulation activation in human endotoxemia.

DETAILED DESCRIPTION:
The beneficial effect of lipid lowering in cardiovascular disease is well established. Statin potently reduce elevated cholesterol levels but also exert pleiotropic other effects such as improvement of inflammation-induced vascular dysfunction, upregulation of endothelial nitric oxide synthase, yield antiinflammatory and antioxidant properties and lower tissue factor (TF) expression on peripheral blood mononuclear cells (PB-MNC) in vivo. The mechanism of action for these effects remains unclear, but is already seen after short term treatment and was independent of cholesterol reduction. Following endotoxin administration to healthy humans, the systemic response includes the activation of inflammation by cytokines, mainly IL-1, IL-6, THF-α and INF-γ, activation of the clotting system with enhanced thrombin generation, and vascular dysfunction, as demonstrable by an impaired response to vasoconstrictors. Low dose endotoxemia therefore serves as an adequate model for acute inflammation and the interaction of the three systems.

The goal of this study is to determine the effect of HMG-CoA reductase inhibitor pretreatment on inflammation and coagulation activation in human endotoxemia and to investigate if anti-inflammatory effects are similar between two different statins. Further, we plan to study genome-wide effects on the leukocyte transcriptome induced by (i) statin pretreatment, (ii) low-dose endotoxemia, and (iii) the anti-inflammatory effects if the statins.

The study will be carried out as a randomized placebo controlled double-blind threeway crossover three period study. Subjects will receive three treatment periods (Day 1 - Day 5) in randomized order consisting of 5 days oral Simvastatin (80 mg/day), 5 days oral Rosuvastatin (40 mg/day) and 5 days adequate placebo. On Day 5 of each study period, subjects will receive LPS (2 ng/kg i.v.). Inflammatory protein expression and coagulation activation will be assessed on Day 1 and Day 5 of each period. Washout-time between treatment periods will be ≥6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 45 years
* Nonsmokers or smokers <5 cig/d
* Body mass index between 18 and 30; respectively weight ≤ 95 kilograms
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Evidence of hypertension, pathologic hyperglycemia, hyperlipidemia
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Start 2006-03; Study Completion 2006-07

PRIMARY OUTCOMES:
monocyte CRP production
leukocyte mRNA expression profiles (human genome GeneChip arrays)

SECONDARY OUTCOMES:
various inflammation and coagulation parameters
platelets
endothelial progenitor cells
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dept. of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Background] Steiner S, Speidl WS, Pleiner J, Seidinger D, Zorn G, Kaun C, Wojta J, Huber K, Minar E, Wolzt M, Kopp CW. Simvastatin blunts endotoxin-induced tissue factor in vivo. Circulation. 2005 Apr 12;111(14):1841-6. doi: 10.1161/01.CIR.0000158665.27783.0C. PMID 15824212
- [Background] Pernerstorfer T, Hollenstein U, Hansen J, Knechtelsdorfer M, Stohlawetz P, Graninger W, Eichler HG, Speiser W, Jilma B. Heparin blunts endotoxin-induced coagulation activation. Circulation. 1999 Dec 21-28;100(25):2485-90. doi: 10.1161/01.cir.100.25.2485. PMID 10604885
- [Derived] Spiel AO, Mayr FB, Leitner JM, Firbas C, Sieghart W, Jilma B. Simvastatin and rosuvastatin mobilize Endothelial Progenitor Cells but do not prevent their acute decrease during systemic inflammation. Thromb Res. 2008;123(1):108-13. doi: 10.1016/j.thromres.2008.03.007. Epub 2008 Apr 22. PMID 18433844